CLINICAL TRIAL: NCT05070130
Title: OpSens dPR for Physiological Assessment of Intermediate Coronary Lesions in Aortic Stenosis
Brief Title: OpSens PRIME CLASS
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: Opsens, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRIME CLASS
Record Dates: First submitted 2021-09-02; First posted 2021-10-07 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Aortic Stenosis
Keywords: Fractional flow reserve; Diastolic pressure ratio; Transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dPR and FFR: Subjects with aortic stenosis who are considered for TAVR will undergo a physiological assessment and prediction of ischemic coronary lesions pre- and post-TAVR by using Opsens non-hyperemic dPR and/or Opsens FFR
  Interventions: Device: dPR and FFR

INTERVENTIONS:
Device: dPR and FFR — OpSens non-hyperemic dPR and/or OpSens FFR

SUMMARY:
In this study it is aimed to determine the diagnostic value of physiological measurements in the presence of aortic stenosis, and whether these are more accurate than angiographic assessment. Post-TAVR FFR will be taken as the reference for predicting ischemic lesions, and angiography and physiology - FFR and diastolic pressure ratio (dPR) - will be performed immediately before and after TAVR, in an all-comer multicentric observational study.

DETAILED DESCRIPTION:
This is a post-marketing, prospective, observational, single arm, multi-center, single country study in Subjects who have severe symptomatic aortic stenosis with a formal indication for TAVR, and one or more intermediate coronary lesions in a relevant coronary artery (>2mm). This study aims to assess if OpSens non-hyperemic dPR (based on a proprietary algorithm) and/or OpSens FFR are suitable methods for the physiological assessment and prediction of ischemic coronary lesions in Subjects with aortic stenosis who are considered for TAVR. This will be done by comparing pre-TAVR measurements of angiography, dPR and FFR and placing them against the post-TAVR FFR, which is considered as the gold standard. Also the post TAVR dPR will be compared with post-TAVR FFR.

A maximum of 137 subjects will be enrolled in 5 to 10 sites in Spain to obtain the required minimum of 137 lesions (see section 11.2 Sample Size Determination) The main hypothesis is that the specificity to predict ischemic lesions in TAVR candidates based on a pre-TAVR dPR ≤ 0.89 is superior compared to the specificity based on angiography alone (both QCA and visual assessment of the stenosis >50%), taking the post-TAVR FFR value of ≤ 0.80 as a reference for positive lesions.

The pressure guidewire used to measure dPR and FFR during diagnostic angiography is the commercially available (CE-marketed) OptoWire family of pressure guidewires from OpSens Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject has a degenerative aortic stenosis with mean valvular gradient ≥40 mmHg
* Subject has a formal heart-team indication for TAVR
* Subject has one or more stable coronary stenosis lesions 30-90% by visual estimation, in a vessel over 2 mm in diameter, and which is amenable for pressure-wire analysis
* Subject agrees to participate in the study and is able to sign the informed consent form

Exclusion Criteria:

* Subject is unable to provide informed consent
* Subject has asthma or acute bronchospasm
* Subject has unstable angina or myocardial infarction
* Subject meets any contraindication in the applicable OptoWire IFU
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have severe symptomatic aortic stenosis with a formal indication for TAVR, and one or more intermediate coronary lesions in a relevant coronary artery (>2mm) are considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Difference between preTAVR dPR specificity and angiography specificity for ischemia | Immediately upon completion of the TAVR procedure
  The difference between PreTAVR dPR specificity (%) - angiography specificity (%), taking post-TAVR FFR as the reference measure.
Diagnostic accuracy | Immediately upon completion of the TAVR procedure
  Establish sufficiently precise estimates (+/- 6.5% around estimate) for the diagnostic accuracy of pre-TAVR dPR expressed in terms of sensitivity and specificity, taking as the reference for ischemia the post-TAVR FFR

SECONDARY OUTCOMES:
Difference in accuracy between dPR and angiography | Immediately upon completion of the TAVR procedure
  The difference between the percentage of lesions correctly classified by preTAVR dPR and the percentage of lesions correctly classified by angiography, always taking postTAVR FFR as the reference measure.
Difference in sensitivity between dPR and angiography | Immediately upon completion of the TAVR procedure
  The difference between the sensitivity of preTAVR dPR and the sensitivity of angiography, where:
  1. preTAVR sensitivity= preTAVR True positive/ (preTAVR true positive+ preTAVR false negative) * 100
  2. angiography sensitivity= angiography True positive/ (angiography true positive+ angiography false negative) * 100,
  taking post-TAVR FFR as the reference measure.
Predicting post-TAVR FFR by pre-TAVR FFR | Immediately upon completion of the TAVR procedure
  Overall diagnostic accuracy of preTAVR FFR, defined as the percentage of lesions correctly classified by pre-TAVR FFR, taking postTAVR FFR as the reference measure.
Difference in accuracy between preTAVR dPR and preTAVR FFR | Immediately upon completion of the TAVR procedure
  The difference in the overall diagnostic accuracy of pre-TAVR dPR and pre-TAVR FFR to predict a post-TAVR FFR ≤ 0.80
Predicting post-TAVR FFR by pre-TAVR hybrid dPR-FFR | Immediately upon completion of the TAVR procedure
  Overall diagnostic accuracyof a pre-TAVR hybrid dPR-FFR based approach to predict a post-TAVR FFR ≤ 0.80

OTHER OUTCOMES:
Success rate | Immediately upon completion of the TAVR procedure
  The success rate of the dPR & FFR procedure, defined as the percentage of cases in which dPR and FFR could be measured, and no procedural complications occurred
Freedom from adenosine administration | Immediately upon completion of the TAVR procedure
  The percentage of Subjects who can be spared the administration of adenosine by a hybrid dPR-FFR strategy, while maintaining an overall diagnostic accuracy ≥ 90%
Percentage of concordance and mean difference between pre- and post-TAVR dPR | Immediately upon completion of the TAVR procedure
  Percentage of concordance and mean difference between pre- and post-TAVR dPR
Percentage of concordance and mean difference between pre- and post-TAVR FFR | Immediately upon completion of the TAVR procedure
  Percentage of concordance and mean difference between pre- and post-TAVR FFR

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Gutierrez Ibanes, MD, Principal Investigator — Hospital Gregoio Maranon
Locations (5):
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Gregorio Maranon, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clinico de Santiago, Santiago de Compostela
  - Hospital Clinico Universitario de Valladolid, Valladolid